CLINICAL TRIAL: NCT06539221
Title: Sphingomyelin in Asthma Pathogenesis
Brief Title: Sphingolipids in Asthma Pathogenesis
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023075
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: asthma; Th17; T-cell senescence; Sphingolipids; ceramide
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate the relationship between the small molecule metabolite sphingolipids and asthma clinical features and explore its involvement in asthma pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* 1. clinical diagnosis of asthma

Exclusion Criteria:

* 1. Combined with chronic obstructive pulmonary disease, bronchiectasis, pneumonia, obstructive sleep apnea hypopnea syndrome, malignant tumor 2. Combined with acute and chronic respiratory failure 3. Combined with severe cardiovascular disease 4. Pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with asthma who visited or were hospitalized in the Department of Respiratory and Critical Care Medicine of Peking University Third Hospital, who met the asthma diagnostic criteria proposed in the Bronchial Asthma Prevention and Treatment Guidelines and healthy controls without history or symptoms of chronic respiratory disease, allergic status or other conditions that could affect the outcome.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
lipidomics | Day 1
  collect blood for lipidomic analysis and in vitro assays

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided